CLINICAL TRIAL: NCT01442948
Title: CD16+ Monocytes in Patients With Coronary Heart Disease
Brief Title: CD16+ Monocytes in Coronary Heart Disease (CHD)
Acronym: PHAMOS
Status: Completed | Type: Observational
Sponsor: Martin-Luther-Universität Halle-Wittenberg (Other)
Responsible Party: Principal Investigator, Axel Schlitt, Senior Physician, Martin-Luther-Universität Halle-Wittenberg
Other Study IDs: CD16PHAMOS
Record Dates: First submitted 2011-09-22; First posted 2011-09-29 (Estimated); Last update posted 2011-09-29 (Estimated); Status verified 2011-09

CONDITIONS: Coronary Heart Disease
Keywords: -CD16+ monocytes
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Acute coronary syndrome
- Stable Angina

SUMMARY:
Monocytes may be separated into phenotypically and functionally distinct cell types by the presence or absence of the lipopolysaccharide receptor CD14 and the Fcγ-receptor CD16. The investigators hypothesize that the total numbers of CD16+ monocytes are significantly related to cardiovascular outcome in patients with angiographically proven coronary heart disease.

ELIGIBILITY:
Inclusion Criteria:

* angiographically proven coronary heart disease
* Age > 18 years

Exclusion Criteria:

* life expectancy < 12 months
* inability to participate in the trial (to give written informed consent)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with angiographically proven coronary heart disease, admitted to the Department of Medicine or Department of Cardiothoracic Surgery of the Martin Luther-University Halle-Wittenberg
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2007-05; Primary Completion 2009-08 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Absolute numbers of CD16+ monocytes stratified by tertiles related to the incidence of the combined endpoint | 12 months
  Incidence of the combined endpoint (non-fatal myocardial infarction, cardiovascular death, stroke) during a follow-up of 12 months

SECONDARY OUTCOMES:
Absolute numbers of CD16+ monocytes stratified by tertiles related to the incidence of each part of the combined endpoint + total death | 12 months
  * non-fatal myocardial infarction
  * cardiovascular death
  * stroke
  * total death
Subgroup analysis for absolute numbers of CD16+ monocytes stratified by tertiles in relation to the combined endpoint | 12 months
  Subgroups of patients:
  Patients with stable Angina Patients with acute coronary syndrome

CONTACTS AND LOCATIONS:
Locations (1):
- University Clinic of the Martin Luther-University Halle-Wittenberg, Halle, Please Select, Germany